CLINICAL TRIAL: NCT00833443
Title: Pharmacogenomics and Medication Development for Methamphetamine Dependence
Brief Title: Study of Medical Treatment for Methamphetamine Addiction
Acronym: BUP PGx
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Keith Heinzerling, Assistant Clinical Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KH_K23; P50DA018185 (NIH); K23DA023558 (NIH); DPMC (Other: NIH / NIDA)
Record Dates: First submitted 2009-01-30; First posted 2009-02-02 (Estimated); Results first posted 2014-02-26 (Estimated); Last update posted 2014-02-26 (Estimated); Status verified 2014-01

CONDITIONS: Methamphetamine; Amphetamine Dependence; Pharmacogenetics; Methamphetamine Dependence; Substance Abuse
Keywords: Methamphetamine; Addiction; Pharmacogenomics; Amphetamine; Bupropion; Meth; Crank; Crystal
MeSH Terms: conditions — Amphetamine-Related Disorders; Substance-Related Disorders; Behavior, Addictive | interventions — Bupropion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bupropion (Active Comparator): Bupropion dose will start at 150 mg per day (one 150 mg sustained release tablet per day) for days 1-3 of the first week. The dose will then be increased to 300 mg per day (one 150 mg sustained release tablet twice daily) on day 4 and will remain 300 mg per day until the last week of the medication phase, when the dose will be decreased to 150 mg per day (one 150 mg sustained release tablet per day) for the last three days.
  Interventions: Drug: Bupropion
- Sugar Pill (Placebo Comparator)
  Interventions: Drug: Bupropion

INTERVENTIONS:
Drug: Bupropion — Bupropion dose will start at 150 mg per day (one 150 mg sustained release tablet per day) for days 1-3 of the first week. The dose will then be increased to 300 mg per day (one 150 mg sustained release tablet twice daily) on day 4 and will remain 300 mg per day until the last week of the medication phase, when the dose will be decreased to 150 mg per day (one 150 mg sustained release tablet per day) for the last three days. The medication treatment phase is for 12 weeks.
  Other Names: Zyban; Wellbutrin

SUMMARY:
Currently there are no medications approved for the treatment of methamphetamine addiction. Bupropion is an antidepressant that is approved by the Food and Drug Administration (FDA) for the treatment of depression and for cigarette smoking cessation but is not approved by the FDA for the treatment of methamphetamine addiction. Preliminary research studies suggest that bupropion may help people receiving treatment for methamphetamine addiction to reduce or to stop their methamphetamine use. But results of these studies also suggest that bupropion may help certain groups of patients more than others, such as men versus women and light versus heavy methamphetamine users, although the reasons for this difference are not known. One possibility is that a person's genetic make up may influence whether or not they respond to treatment with bupropion for methamphetamine addiction.

The purpose of the study is to determine if bupropion is can help people reduce or stop their methamphetamine use and to investigate whether genetic variations influence whether people respond to treatment with bupropion for methamphetamine addiction, which may help doctors and patients better decide if treatment with bupropion will be beneficial or not. To identify possible genetic variations that influence response to bupropion, we will perform genetic tests on blood or saliva specimens from participants receiving treatment with either bupropion or placebo (which is a pill that contains no medication) in conjunction with standard cognitive behavioral therapy drug counseling. We will compare methamphetamine use, as assessed with urine drug screens, among participants receiving bupropion versus those receiving placebo to determine if bupropion helps people to reduce or stop their methamphetamine use. We will then compare the results of the genetic tests among participants who respond and who do not respond to bupropion. In addition, since the amount of methamphetamine a person uses was associated with response to bupropion in preliminary studies, we will also compare the results of genetic testing among persons with heavy versus light methamphetamine use before entering treatment.

Results of this study have the potential to provide insights into the biology of methamphetamine addiction and help increase the understanding of how bupropion works. This information could be useful to develop effective medications for methamphetamine addiction and to improve the ability of clinicians to provide treatment to patients with methamphetamine addiction.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older;
2. meet DSM-IV criteria for methamphetamine dependence;
3. seeking treatment for MA problems;
4. specific range of methamphetamine use in the 30 days prior to study entry;
5. willing and able to comply with study procedures, including genotyping;
6. willing and able to provide written informed consent;
7. if female, not pregnant or lactating and willing to use an acceptable method of barrier birth control (e.g. condoms) during the trial.

Exclusion Criteria:

1. have a medical condition that, in the study physician's judgment, may interfere with safe study participation (e.g., active TB, unstable cardiac, renal, or liver disease, unstable diabetes);
2. have a current neurological disorder (e.g., organic brain disease, dementia) or major psychiatric disorder not due to substance abuse (e.g., schizophrenia, bipolar disorder) as assessed by the SCID or a medical history which would make study agent compliance difficult or which would compromise informed consent, or recent (past 30 days) history of suicide attempts and/or current serious suicidal intention or plan as assessed by the SCID;
3. currently on prescription medication that is contraindicated for use with bupropion;
4. have current dependence on cocaine, opiates, alcohol, or benzodiazepines as defined by DSM-IV-TR;
5. have a history of alcohol dependence within the past three years;
6. have a history of a seizure disorder;
7. have a medical condition (such as serious head injury) that is associated with increased risk of seizures or on a medication that lowers the seizure threshold;
8. have a history of anorexia or bulimia;
9. have current hypertension uncontrolled by medication, or any other circumstances that, in the opinion of the investigators, would compromise participant safety;
10. have a history of sensitivity to bupropion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2009-01; Primary Completion 2012-12 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keith G Heinzerling, MD MPH, Principal Investigator — UCLA Dept of Family Medicine
Locations (1):
- UCLA Clinical Research Site 910 Vine St, Los Angeles, California, United States

REFERENCES:
- [Derived] Heinzerling KG, Swanson AN, Hall TM, Yi Y, Wu Y, Shoptaw SJ. Randomized, placebo-controlled trial of bupropion in methamphetamine-dependent participants with less than daily methamphetamine use. Addiction. 2014 Nov;109(11):1878-86. doi: 10.1111/add.12636. Epub 2014 Aug 5. PMID 24894963

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited via advertisements and outreach in the Los Angeles area
Period: Overall Study
Arm/Group | Bupropion | Sugar Pill
Started | 41 | 43
Completed | 21 | 15
Not Completed | 20 | 28

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bupropion | Sugar Pill | Total
Number analyzed (Participants) | 41 | 43 | 84
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.6 (10.1) | 38.1 (10.3) | 38.4 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 9 | 16
  Male | 34 | 34 | 68
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic | 18 | 17 | 35
  White | 15 | 13 | 28
  African American | 7 | 10 | 17
  Asian/Pacific Islander | 1 | 3 | 4
Region of Enrollment [Number; unit: participants]
  United States | 41 | 43 | 84

OUTCOME MEASURES:

1. Primary Outcome: Treatment Effectiveness Score
Description: The mean number of methamphetamine-free urine drug screens provided by participants in each group (range 0-36)
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: urine drug screens
Arm/Group | Bupropion | Sugar Pill
Number analyzed (Participants) | 41 | 43
urine drug screens | 16.1 (12.7) | 10.6 (11.2)

2. Primary Outcome: End of Treatment Methamphetamine Abstinence
Description: Methamphetamine abstinence confirmed via urine drug screens during the final two weeks of treatment (weeks 11 and 12)
Time Frame: 12 weeks
Measure: Number; unit: participants
Arm/Group | Bupropion | Sugar Pill
Number analyzed (Participants) | 41 | 43
participants | 12 | 6

3. Secondary Outcome: Treatment Retention
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Bupropion | Sugar Pill
Number analyzed (Participants) | 41 | 43
days | 61.0 (28.8) | 49.5 (31.7)

4. Post Hoc Outcome: End of Treatment Methamphetamine Abstinence
Time Frame: 12 weeks
Measure: Number; unit: participants
Groups:
- Medication Adherent: Participants in the bupropion group with a week 6 bupropion/hydroxybupropion plasma levels suggesting medication adherence
- NOT Medication Adherent: Participants in the bupropion group with a week 6 bupropion/hydroxybupropion plasma levels suggesting medication NON-adherence
Arm/Group | Medication Adherent | NOT Medication Adherent
Number analyzed (Participants) | 13 | 28
participants | 7 | 5

ADVERSE EVENTS:
Arm/Group | Bupropion | Sugar Pill
Serious Adverse Events (participants affected / at risk) | 2/41 | 2/43
Other Adverse Events (participants affected / at risk) | 29/41 | 17/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bupropion (N=41) | Sugar Pill (N=43)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 1 (1)
Chest pain (Cardiac disorders) | 1 (1) | 0 (0)
Liver abscess (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bupropion (N=41) | Sugar Pill (N=43)
Insomnia (Psychiatric disorders) | 9 | 6
"Amped up" (Psychiatric disorders) | 6 | 2
Depressed mood (Psychiatric disorders) | 5 | 3
Headache (Nervous system disorders) | 5 | 1
Diarrhea (Gastrointestinal disorders) | 4 | 0
Dry mouth (Gastrointestinal disorders) | 3 | 2
Nausea/vomiting (Gastrointestinal disorders) | 3 | 1
Dizziness (Nervous system disorders) | 2 | 1
Elevated blood pressure (Cardiac disorders) | 2 | 0
Muscle twitching (Nervous system disorders) | 2 | 0
Panic attack (Psychiatric disorders) | 2 | 1
Paranoia (Psychiatric disorders) | 2 | 0
Vivid dreams/nightmares (Psychiatric disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No